CLINICAL TRIAL: NCT01647217
Title: Safety and Efficacy of Single-use Terpinen-4-ol Pads for Treating Ocular Mites A Randomized Clinical Trial
Brief Title: Demodex Blepharitis Treatment Study
Acronym: DBTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P012-01; 2R44EY019586-02 (NIH)
Record Dates: First submitted 2012-07-12; First posted 2012-07-23 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-05

CONDITIONS: Chronic Blepharitis
Keywords: Blepharitis; Demodex; Mites; Tea Tree oil; Terpinen
MeSH Terms: conditions — Blepharitis | interventions — terpinenol-4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terpinen-4-ol Treatment Arm (Experimental): 8 patients will be randomized into the Study Group and will be subdivided into 2 subgroups (3 / 5 patients) according to the treatment regimen (once or twice per day). Changes in the mite counts will be correlated with changes in symptoms and signs.
  Interventions: Drug: Terpinen-4-ol
- Placepo Pads Contol Arm (Placebo Comparator): 9 patients will be randomized into the control group and will be treated with placebo pads. They will be divided into 2 subgroups (5 / 4 patients) according to the frequency (once or twice per day). Changes in the mite counts will be correlated with changes in symptoms and signs.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Terpinen-4-ol — Lid scrub once or twice per day for one month.
  Other Names: T4O
  Arms: Terpinen-4-ol Treatment Arm
Other: Placebo — Lid scrub once or twice per day for one month
  Arms: Placepo Pads Contol Arm

SUMMARY:
This is a randomized clinical trial to determine the safety and efficacy of terpinen-4-ol (T4O), the most active ingredient of tea tree oil (TTO), in eradicating ocular demodicosis (reducing ocular demodex counts and achieving the clinical improvement with minimal or no irritation).

DETAILED DESCRIPTION:
Demodex blepharitis is one of the most common causes of chronic blepharitis. The investigators preliminary clinical study showed that lid scrub with TTO was effective in resolving chronic blepharoconjunctivitis; however, it was not convenient for self-administration and caused irritation in some patients. Preclinical safety studies have verified that T4O is less irritant. In this study, the investigators will determine the optimal regimen of T4O Pads.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Demodex blepharitis for duration of at least 3 months.
* Age range: 15-80 years old.
* Both genders and all ethnic groups comparable with the local community.
* Able to understand and willing to sign a written informed consent
* Able and willing to cooperate with the investigational plan.
* Able and willing to complete all mandatory follow-up visits.

Exclusion Criteria:

* Patients who are currently engaged in another clinical trial, unwilling or unable to give consent, to accept randomization, or to return for scheduled visits.
* Children under 15.
* Pregnant women or expecting to be pregnant during the study.
* Systemic immune deficient conditions such as AIDS or under systemic immunosuppressant.
* Concomitant use of ophthalmic topical medications (excluding non-preserved tear substitutes).
* Concomitant use of systemic antibiotics or steroids.
* Contact lens wear (unless discontinued for ≥ 30 days before randomization)
* Active ocular infection or allergy
* Unable to close eyes or uncontrolled blinking
* Presence of aqueous tear deficient dry eye defined by the Fluorescein Clearance Test as less than 3 mm wetting in 1-minute Schirmer test with anesthesia.
* Previous allergic reaction to TTO-containing products or cosmetic fragrance.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scheffer CG Tseng, MD, PhD, Study Chair — BioTissue Holdings, Inc
Locations (1):
- Ocular Surface Center, Miami, Florida, United States

REFERENCES:
- [Background] Gao YY, Di Pascuale MA, Li W, Liu DT, Baradaran-Rafii A, Elizondo A, Kawakita T, Raju VK, Tseng SC. High prevalence of Demodex in eyelashes with cylindrical dandruff. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3089-94. doi: 10.1167/iovs.05-0275. PMID 16123406
- [Background] Gao YY, Di Pascuale MA, Li W, Baradaran-Rafii A, Elizondo A, Kuo CL, Raju VK, Tseng SC. In vitro and in vivo killing of ocular Demodex by tea tree oil. Br J Ophthalmol. 2005 Nov;89(11):1468-73. doi: 10.1136/bjo.2005.072363. PMID 16234455
- [Background] Gao YY, Di Pascuale MA, Elizondo A, Tseng SC. Clinical treatment of ocular demodecosis by lid scrub with tea tree oil. Cornea. 2007 Feb;26(2):136-43. doi: 10.1097/01.ico.0000244870.62384.79. PMID 17251800
- [Background] Kheirkhah A, Casas V, Li W, Raju VK, Tseng SC. Corneal manifestations of ocular demodex infestation. Am J Ophthalmol. 2007 May;143(5):743-749. doi: 10.1016/j.ajo.2007.01.054. Epub 2007 Mar 21. PMID 17376393
- [Background] Kheirkhah A, Blanco G, Casas V, Tseng SC. Fluorescein dye improves microscopic evaluation and counting of demodex in blepharitis with cylindrical dandruff. Cornea. 2007 Jul;26(6):697-700. doi: 10.1097/ICO.0b013e31805b7eaf. PMID 17592319
- [Background] Li J, O'Reilly N, Sheha H, Katz R, Raju VK, Kavanagh K, Tseng SC. Correlation between ocular Demodex infestation and serum immunoreactivity to Bacillus proteins in patients with Facial rosacea. Ophthalmology. 2010 May;117(5):870-877.e1. doi: 10.1016/j.ophtha.2009.09.057. Epub 2010 Jan 15. PMID 20079929
- [Background] Liang L, Safran S, Gao Y, Sheha H, Raju VK, Tseng SC. Ocular demodicosis as a potential cause of pediatric blepharoconjunctivitis. Cornea. 2010 Dec;29(12):1386-91. doi: 10.1097/ICO.0b013e3181e2eac5. PMID 20847679
- [Background] Liu J, Sheha H, Tseng SC. Pathogenic role of Demodex mites in blepharitis. Curr Opin Allergy Clin Immunol. 2010 Oct;10(5):505-10. doi: 10.1097/ACI.0b013e32833df9f4. PMID 20689407
- [Background] Gao YY, Xu DL, Huang lJ, Wang R, Tseng SC. Treatment of ocular itching associated with ocular demodicosis by 5% tea tree oil ointment. Cornea. 2012 Jan;31(1):14-7. doi: 10.1097/ICO.0b013e31820ce56c. PMID 21955627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Terpinen-4-ol Treatment Arm | Placepo Pads Contol Arm
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terpinen-4-ol Treatment Arm | Placepo Pads Contol Arm | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (21.2) | 49 (18.5) | 48.8 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Demodex Mites
Description: Change in mites count after treatment compared to the baseline data. If the mites' count remains zero during the last two visits, it is considered "complete eradication". Patients without achieving complete eradication will be categorized as "incomplete eradication".
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Mites
Groups:
- Terpinen-4-ol Treatment Arm: 10 patients will be randomized into the Study Group and will be subdivided into 2 subgroups (5 patients each) according to the treatment regimen (once or twice per day). Changes in the mite counts will be correlated with changes in symptoms and signs.
  Terpinen-4-ol: Lid scrub once or twice per day for one month.
- Placepo Pads Contol Arm: 10 patients will be randomized into the control group and will be treated with placebo pads. They will be divided into 2 subgroups (5 each) according to the frequency (once or twice per day). Changes in the mite counts will be correlated with changes in symptoms and signs.
  Placebo: Lid scrub once or twice per day for one month
Arm/Group | Terpinen-4-ol Treatment Arm | Placepo Pads Contol Arm
Number analyzed (Participants) | 7 | 8
Mites | -3 (3.1) | -0.4 (3.6)

2. Secondary Outcome: Change in Lid Margin Redness and Bulbar Conjunctival Hyperemia
Description: Lid margin redness and bulbar conjunctival hyperemia were each assessed using an ordered categorical value ranging from 0 (None) to 3 (Severe). The two scores were summed to obtain the final score, which ranges from 0 (None) to 6 (Severe).
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Terpinen-4-ol Treatment Arm | Placepo Pads Contol Arm
Number analyzed (Participants) | 7 | 8
units on a scale | -2.3 (1.4) | -3.1 (1.9)

ADVERSE EVENTS:
Arm/Group | Terpinen-4-ol Treatment Arm | Placepo Pads Contol Arm
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes